CLINICAL TRIAL: NCT00130429
Title: Phase II Randomised, Double Blind, Placebo Controlled, Parallel Group Study to Investigate the Safety, Effect on Cognition and Pharmacokinetic Profile of PYM50028 in Subjects With Mild Dementia of the Alzheimer's Type
Brief Title: Safety and Effect on Memory of PYM50028 in Mild Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phytopharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P58/09ME/03/04
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Alzheimer's Disease
Keywords: dementia; memory; Hopkins verbal learning test; paired associated learning
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — sarsasapogenin

INTERVENTIONS:
Drug: PYM50028

SUMMARY:
The purpose of this study is to assess the effect of PYM50028 administered once daily for up to 12 weeks on the memory and other faculties of subjects with dementia due to Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* At least 50 years of age
* Diagnosis of possible or probable Alzheimer's disease
* Mini mental state examination score at least 16
* Good understanding of both written and verbal English
* A recent head scan that is consistent with the diagnosis of Alzheimer's disease

Exclusion Criteria:

* Recent history or clinical evidence of significant neurological disease other than dementia due to Alzheimer's disease
* Known to have another condition that is associated with dementia
* Use of psychotropic medication within the previous 4 weeks (excluding cholinesterase inhibitors, selective serotonin reuptake inhibitors and venlafaxine)
* Hormone replacement therapy started or changed within the previous 6 months
* Received any investigational drugs within the previous 12 weeks

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2004-01; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Hopkins verbal learning test (revised) total word recall after 12 weeks
Cambridge neuropsychological test automated battery (CANTAB) paired associate learning (Phytopharm modified form) total adjusted error score after 12 weeks

SECONDARY OUTCOMES:
Mini mental state examination score
Clinical dementia rating (overall and sum of boxes)
CANTAB rapid visual information processing (RVIP) mean latency
CANTAB RVIP total correct hits
CANTAB spatial working memory within error, between error and strategy scores
Clinicians global impression of change
Disability assessment for dementia score

CONTACTS AND LOCATIONS:
Overall Officials: Robin Jacoby, FRCPsych, Principal Investigator — University of Oxford, UK
Locations (1):
- Oxford Project to Investigate Memory and Ageing, Oxford, Oxfordshire, United Kingdom